CLINICAL TRIAL: NCT04071002
Title: Functional Status and Activity Participation Levels in Patients With Distal Radius Fracture
Brief Title: Patients With Distal Radius Fracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, HANDE USTA, Principal Investigator, Research Assistant, Pamukkale University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3518
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Physical Disability
Keywords: Distal radius fracture; functional status; activity participation; hand therapy
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- surgical group (Active Comparator): distal radius fractures that treated volar plate
  Interventions: Other: 12 weeks physical therapy programme
- conservative group (Active Comparator): distal radius fractures that treated plaster of paris
  Interventions: Other: 12 weeks physical therapy programme

INTERVENTIONS:
Other: 12 weeks physical therapy programme — The programme include contrast bath, bandage, massage, active exercises, resistive exercises.

SUMMARY:
Surgically and conservatively treated distal radius fractures followed for six month. In this period 12 weeks rehabilitation programme applied for each group. Nine different evaluations were done in the initial, after physical therapy and 6th month. Results were presented.

DETAILED DESCRIPTION:
Distal radius fracture (DRF) affects overall health status. The International Classification of Function (ICF) based approach is appropriate in the management of DRF. The purpose of this study was to investigate functional status and activity participation levels of DRF patients.

The patients were divided into conservative and surgical groups and were admitted to 12-weeks rehabilitation period. The evaluation of the body function and structure were done with Visual Analogue Scale, algometer, range of motion (ROM) and grip strength. Also, radiographic evaluations were done. Activity participation assessments were done with Push-Off Test (POT), Michigan Hand Outcomes Questionnaire (MHOQ), Short Form of Disabilities of Arm-Shoulder and Hand Questionnaire (Q-DASH) and Jebsen-Taylor Hand Function Test (JTHFT). Mann-Whitney U and Wilcoxon Tests were used respectively for intergroup and intra-group comparisons. Statistical significance level was p<0,05.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 60
* Diagnosed with distal radius fracture
* Primary fixation after injury.

Exclusion Criteria:

* Bilateral distal radius fracture
* Concomitant ulna styloid fracture
* Another orthopaedic, neurological or rheumatologic problem involving the ipsilateral upper limb
* Patients who underwent surgery that involved ipsilateral upper extremity
* Associated injuries such as nerve or tendon injuries
* Secondary procedures at follow-up
* Un-cooperated patients.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2015-01-21 (Actual); Primary Completion 2016-06-09 (Actual); Study Completion 2016-09-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | six month
  To evaluate pain severity, patient show a point to indicate her/his pain between 0-10 points on a vertical 100mm line. Severity of pain was assessed with VAS in sleep, rest, and activity.
algometer | six month
  An algometer is used to evaluate pain threshold of the patient for distal radioulnar joint, ulnas styloid, m.pronator quadratus, radial styloid, m. flexor pollicis longus, and triangular fibrocartilage complex.The threshold value of pain was recorded by placing the probe against the points. Then, it was gradually increased and reduced to apply a pressure of 1kg / 0.5cm² with 0.5 cm² probe head .
range of motion | six month
  An universal goniometer is used to evaluate patient's active motion of joints for wrist and forearm.
grip strength | six month
  Grip strength was measured by a hand dynamometer according to the American Association of Hand Therapy Association's standard grip strength measurement method. Right/left extremity and their progression are compared in this evaluation.
radiographic evaluations | six month
  The posteroanterior (PA) and lateral (L) radiographic measurements were assessed by an experienced hand surgeon to determine the type of fracture, geometry, and associated pathology. Radial length and radial inclination were assessed by PA radiography. Dorsal or volar angulations of the distal fragment were evaluated on the lateral radiography.
Push-Off Test (POT) | six month
  POT was performed to determine the weight transfer strength of the patient to the injured extremity. The test was performed simultaneously and bilaterally by reversing the hand parts of the two hand dynamometers.
Michigan Hand Outcomes Questionnaire (MHOQ) | six month
  MHOQ was used for evaluating the participation and functional levels of the patients. In the questionnaire consisting of 37 questions under six headings, general hand function, daily life activities, pain, work, aesthetics and satisfaction are evaluated. In the pain scale, high scores indicate greater pain, while in the other five scales, high scores denote better hand performance.
Short Form of Disabilities of Arm-Shoulder and Hand Questionnaire (Q-DASH) | six month
  It was used to assess the upper extremity functional status of patients from their perspective. It is a questionnaire that measures an individual's ability to complete tasks, absorb forces, and severity of symptoms. It includes 11 item. The score on test ranges from 0 (no disability) to 100 (most severe disability). A higher scores indicate a greater level of disability and severity.
Jebsen-Taylor Hand Function Test (JTHFT) | six month
  The seven individual subtests of JTHFT writing, card turning, picking up small common objects, stacking checkers, stimulated feeding, moving light objects and moving heavy objects, were performed as a standardized procedure.

CONTACTS AND LOCATIONS:
Overall Officials: HANDE USTA, MSC, Principal Investigator — Pamukkale University; ALI KITIS, PROF, Study Chair — Pamukkale University; AHMET FAHIR DEMIRKAN, PROF, Study Director — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Kinikli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Valdes K, Naughton N, Michlovitz S. Therapist supervised clinic-based therapy versus instruction in a home program following distal radius fracture: a systematic review. J Hand Ther. 2014 Jul-Sep;27(3):165-73; quiz 174. doi: 10.1016/j.jht.2013.12.010. Epub 2014 Jan 3. PMID 24508093